CLINICAL TRIAL: NCT05006794
Title: A Phase 1a/b Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GS-9716 as Monotherapy and in Combination With Anticancer Therapies in Subjects With Solid Malignancies
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GS-9716 as Monotherapy and in Combination With Anticancer Therapies in Adults With Solid Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-467-5643
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Solid Malignancies
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: zamzetoclax Dose-Escalation (Experimental): Patients will receive escalating doses of zamzetoclax to estimate MTD.
  Interventions: Drug: zamzetoclax
- Part A: zamzetoclax Dose-Expansion (Experimental): Patients will receive ≤ MTD of zamzetoclax.
  Interventions: Drug: zamzetoclax
- Part B (Cohort B1): Zamzetoclax + docetaxel (Experimental): Patients will receive escalating doses of zamzetoclax in combination with docetaxel.
  Interventions: Drug: zamzetoclax; Drug: Docetaxel
- Part B (Cohort B4): zamzetoclax + sacituzumab govitecan-hziy (Experimental): Patients will receive escalating doses of zamzetoclax in combination with sacituzumab govitecan-hziy.
  Interventions: Drug: zamzetoclax; Drug: sacituzumab govitecan-hziy
- Part C (Cohort C1): zamzetoclax + docetaxel (Experimental): Patients will receive ≤ MTD zamzetoclax in combination with docetaxel.
  Interventions: Drug: zamzetoclax; Drug: Docetaxel
- Part C (Cohort C4): zamzetoclax + sacituzumab govitecan-hziy (Experimental): Patients will receive ≤ MTD zamzetoclax in combination with sacituzumab govitecan-hziy.
  Interventions: Drug: zamzetoclax; Drug: sacituzumab govitecan-hziy

INTERVENTIONS:
Drug: zamzetoclax — Tablet(s) administered orally
  Other Names: GS-9716
Drug: Docetaxel — Administered intravenously
  Arms: Part B (Cohort B1): Zamzetoclax + docetaxel; Part C (Cohort C1): zamzetoclax + docetaxel
Drug: sacituzumab govitecan-hziy — Administered intravenously
  Arms: Part B (Cohort B4): zamzetoclax + sacituzumab govitecan-hziy; Part C (Cohort C4): zamzetoclax + sacituzumab govitecan-hziy

SUMMARY:
This is a Phase I open-label, multi-center study of zamzetoclax (formerly GS-9716) tested either as monotherapy or in combination with other anti-cancer agents in patients with advanced solid malignancies. Primary objectives are to define the maximum tolerated dose (MTD) or maximum administered dose of zamzetoclax, and characterize the safety and tolerability of zamzetoclax as monotherapy and in combination with anti-cancer therapies.

ELIGIBILITY:
Key Inclusion Criteria:

General Inclusion Criteria (all cohorts):

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease per RECIST version 1.1
* Adequate hematology, renal and hepatic function
* Left ventricular ejection fraction (LVEF) ≥ 50%
* Patients with brain metastases may be enrolled only if treated, nonprogressive, asymptomatic and not taking high dose steroids for at least 4 weeks prior to Cycle 1 Day 1 (C1D1)
* Individuals of childbearing potential who engage in heterosexual intercourse must agree to use method(s) of contraception, per protocol.
* Tissue criteria: must provide sufficient, and adequate tumor tissue sample or agree to have a biopsy taken.

Part A Specific Inclusion Criteria: zamzetoclax as monotherapy

* Histologically or cytologically confirmed locally advanced or metastatic malignant solid tumor for which no standard therapy is available, standard therapy has failed, or for whom standard-of-care therapy is contraindicated.

Cohorts B1 and C1 Specific Inclusion Criteria:

* Histologically or cytologically confirmed unresectable metastatic or locally advanced disease following treatment for metastatic disease including an immune checkpoint inhibitor and a platinum-containing chemotherapy
* Patients with actionable genomic alterations must have also received treatment with at least 1 approved therapy appropriate to the genomic alteration unless unavailable or contraindicated

Cohorts B4 and C4 Specific Inclusion Criteria:

* Histologically or cytologically confirmed disease based on the most recent analyzed biopsy metastatic disease that is refractory to or relapsed after at least 2 prior standard-of-care chemotherapy regimens, one of which was a taxane (unless contraindicated).

Key Exclusion Criteria:

* Prior systemic anti-cancer therapy must meet wash-out criteria outlined in protocol
* Treatment with any high dose systemic corticosteroids or nonsystemic radiotherapy within 2 weeks of the first dose of zamzetoclax (low dose corticosteroids permitted).
* Women who are pregnant or lactating
* Patients with active ≥ Grade 2 nausea or vomiting, and/or signs of intestinal obstruction
* Known active or chronic hepatitis B or C infection or HIV infection/ HIV positive
* Known history of clinically significant cardiovascular disease or heart failure.
* Known history of clinically significant active chronic obstructive pulmonary disease or other moderate to severe chronic respiratory illness present within 6 months prior to C1D1
* Known history of other clinically significant pulmonary disease or evidence of active pneumonitis
* Uncontrolled pleural effusion, pericardial effusion, or ascites
* History of clinically significant bleeding, intestinal obstruction, or gastrointestinal (GI) perforation within 6 months prior to C1D1
* Infection requiring intravenous anti-infective use within 2 weeks prior to C1D1
* Active or history of autoimmune disease or immune deficiency
* History of uncured coexisting cancer, not including uncured basal cell carcinoma, cervical cancer in situ, or superficial bladder cancer.

Cohort A Specific Exclusion Criteria: zamzetoclax as monotherapy:

* Known heart failure or elevated cardiac biomarkers

Cohorts B1 and C1 Specific Exclusion Criteria:

* Known hypersensitivity to excipients in study treatments.

Cohorts B4 and C4 Specific Exclusion Criteria:

* Prior treatment with sacituzumab govitecan-hziy or a topoisomerase 1 inhibitor or agents targeting Trop-2.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients Experiencing Dose-Limiting Toxicities (DLTs) | First dose date up to 28 days
Percentage of Patients Experiencing Adverse Events (AEs) According to National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE), Version 5.0 | First dose date up to last dose date (Maximum: 105 weeks) plus 30 days

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) for Zamzetoclax | Approximately 105 Weeks
Time to Maximum Observed Concentration (Tmax) for Zamzetoclax | Approximately 105 Weeks
Area Under the Concentration Versus Time Curve From Time 0 to 24 Hours (AUC0-24) for Zamzetoclax | Approximately 105 Weeks
Parts B and C: Objective Response Rate (ORR) | Up to 105 weeks
  ORR is defined as the percentage of patients who achieve a confirmed complete response (CR) or confirmed partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Parts B and C: Disease Control Rate (DCR) | Up to 105 weeks
  DCR is defined as the percentage of patients who achieve a CR, PR, or stable disease (SD) as assessed by RECIST version 1.1.
Parts B and C: Progression-Free Survival (PFS) | First dose date to PD or death, whichever occurs first (up to 39 months)
  PFS is defined as the interval from the first dose of zamzetoclax to the earlier of the first documentation of definitive progressive disease (PD) or death from any cause.
Parts B and C: Time to Response (TTR) | First dose date to the first documentation of CR or PR (up to 105 weeks)
  TTR is defined as the time from first dose of zamzetoclax to the first documentation of CR or PR.
Parts B and C: Duration of Response (DOR) | From first documentation of CR or PR to PD or death, whichever occurs first (up to 37 months)
  DOR is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of definitive disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (13):
- United States (10):
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - START Midwest, Grand Rapids, Michigan
  - Montefiore Medial Center - Montefiore Medical Park, The Bronx, New York
  - Novant Health Cancer Institute - Elizabeth (Breast Cancer), Charlotte, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health Oregon Health & Sciences University-Knight Cancer Institute, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center- Ein Kerem, Jerusalem
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-467-5643